CLINICAL TRIAL: NCT07017660
Title: Effect of Virtual Reality Application on Pain, Anxiety and Patient Satisfaction During Cystoscopy: A Randomized Controlled Trial
Brief Title: Virtual Reality Application During Cystoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayten Akkaya (Other)
Responsible Party: Sponsor-Investigator, Ayten Akkaya, Assist. Prof. Dr., Ankara Medipol University
Organization: Ankara Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-022
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Virtual Reality; Rigid Cystoscopy
Keywords: Cystoscopy; Pain; anxiety; satisfaction; virtual reality
MeSH Terms: conditions — Pain; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): Routine institution procedures will be applied during the cystoscopy procedure.
  Interventions: Other: No intervention
- virtual reality glasses (Experimental): Patients will be asked to wear virtual reality glasses starting three minutes before the procedure and until the procedure is completed. The patient will be shown a video of nature scenes with the virtual reality glasses and will also be made to listen to the sounds of water and birds. Routine institution procedures will be applied during the cystoscopy procedure.
  Interventions: Other: virtual reality glasses

INTERVENTIONS:
Other: virtual reality glasses — Patients will be asked to wear virtual reality glasses starting three minutes before the procedure and until it is completed. With the virtual reality glasses, the patient will be shown a video of nature scenes and made to listen to the sounds of water and birds. Routine institutional procedures will be applied during the cystoscopy procedure.
  Arms: virtual reality glasses
Other: No intervention — Routine institution procedures will be applied during the cystoscopy procedure.
  Arms: control group

SUMMARY:
This randomized controlled experimental study aimed to determine the effect of virtual reality glasses during cystoscopy on pain, anxiety and patient satisfaction.

DETAILED DESCRIPTION:
Patients in the intervention arm; In order to evaluate pain, anxiety and patient satisfaction regarding the cystoscopy procedure, the patient's pain level will be assessed with the Visual Analog Scale 10 minutes before the procedure and the patient's anxiety level will be assessed with the State Anxiety Scale. Patients will be asked to wear virtual reality glasses starting three minutes before the procedure and until the procedure is completed. The patient will be shown a video of nature scenes with the virtual reality glasses and will also be made to listen to the sounds of water and birds. Routine institution procedures will be applied during the cystoscopy procedure. 10 minutes after the procedure, the patient's pain and satisfaction level will be assessed with the Visual Analog Scale and the patient's anxiety level will be assessed with the State Anxiety Scale.

Patients in the control arm; To assess pain, anxiety, and patient satisfaction with the cystoscopy procedure, the patient's pain level will be assessed with the Visual Analog Scale and the patient's anxiety level will be assessed with the State Anxiety Scale 10 minutes before the procedure. Routine institution procedures will be applied during the cystoscopy procedure. 10 minutes after the procedure, the patient's pain and satisfaction levels will be assessed with the Visual Analog Scale and the patient's anxiety level will be assessed with the State Anxiety Scale.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older,
* First elective and rigid cystoscopy performed under local anesthesia,
* No vision, hearing and perception problems,
* Open to communication and able to speak Turkish,
* Patients who agree to participate in the study

Exclusion Criteria:

* Contraindications for the procedure (lidocaine allergy, urinary tract infection, anatomical problems related to the urethra, etc.)
* Use of any analgesic or sedative medication at least 4 hours before cystoscopy Patients who undergo manipulation such as J stent placement or removal and/or bladder biopsy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog scale | 1 day
  Rating is done on a scale with a 10 cm horizontal or vertical ruler and "0" means dissatisfaction and "10" means the highest level of satisfaction.
Visual Analog Scale | 1 day
  Grading is made with a 10 cm long horizantal or vertical ruler on the scale and "0" means no pain and "10" means the most severe pain.
Spielberg State Anxiety Scale | 1 day
  The scale has a four-point Likert structure consisting of 20 items, and a total score of 20-80 is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Ayten Akkaya, PhD, Principal Investigator — Ankara Medipol University Faculty of Health Sciences, Department of Nursing
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No